CLINICAL TRIAL: NCT05475795
Title: Postoperative Pain After Pulpectomy of Primary Molars Using Different Obturation Materials: A Parallel Randomized Clinical Trial
Brief Title: Postoperative Pain After Pulpectomy of Primary Molars Using Different Obturation Materials
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Nada Mohamed Hassan, Postgraduate student at Faculty of Dentistry Minia University, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 576-2022
Record Dates: First submitted 2022-07-24; First posted 2022-07-27 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Metapex; Endoflas F.S.

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metapex group (Active Comparator): Obturation of primary molars with calcium hydroxide and iodoform paste
  Interventions: Other: Metapex; Other: Endoflas
- Endoflas group (Experimental): Obturation of primary molars with calcium hydroxide, eugenol and iodoform paste
  Interventions: Other: Metapex; Other: Endoflas

INTERVENTIONS:
Other: Metapex — obturation of root canals of primary molars with Metapex
Other: Endoflas — obturation of root canals of primary molars with Endoflas

SUMMARY:
Testing postopertive pain after pulpectomy of primary molars with Metapex and Endoflas using modified Wong-Baker scale of pain.

DETAILED DESCRIPTION:
The current equivalent parallel randomized controlled trial will be conducted to evaluate intensity and duration of post-operative pain after pulpectomy of asymptomatic necrotic primary molars, using Metapex and Endoflas obturation materials

ELIGIBILITY:
Inclusion Criteria:

* 3.1. Inclusion criteria: The study will include children who meet the following clinical and radiographic criteria:

Clinical:

1. 5-7-year old children categorized as class I or II according to American Society of Anaesthesiologists (ASA) scale.
2. Children rated as no.3 or 4 in Frankel behavior rating scale (FBRS).
3. Presence of at least one primary molar with deep carious lesion.
4. Asymptomatic necrotic molars confirmed by the absence of bleeding on opening of the pulp chamber.

Radiographic:

1. Extensive caries approaching to the pulp.
2. Presence of at least two-thirds of root length.

Exclusion Criteria:

* A child's tooth with any of the following criteria:

Clinical findings:

1. History of spontaneous unprovoked toothache.
2. Extensive crown destruction that preclude coronal restoration.
3. Presence of adjacent or opposing tooth with deep carious lesion "in the same side".
4. History of administering analgesics 12 hours before tooth obturation.

Radiographic findings:

1. Presence of a large furcation or periapical radiolucency approximating the succedaneous tooth.
2. Presence of pathological internal/external root resorption.
3. Absence of underlying permanent successor.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-01-16 (Estimated)

PRIMARY OUTCOMES:
postoperative pain. | after one day and after one week .
  Measuring post operative pain after pulpectomy with two different obturation materials using (Modified Wong-backer scale of pain )which have four scales from( 0 to 3) which 0 is the better outcome( no pain) and 3 is the worst (severe pain).

CONTACTS AND LOCATIONS:
Overall Officials: Osama S Gad El-Hak, PhD, Study Director — Pediatric Dentistry Department, Faculty of Dentistry, Minia University
Locations (1):
- Nada Mohamed Hassan Saied, Minya, Egypt